CLINICAL TRIAL: NCT04924153
Title: A Non-Drug, Longitudinal, Prospective Natural History Study of Individuals With KCNT1-Related Epilepsy (K1Te)
Brief Title: A Natural History Study of Participants With Potassium Sodium-Activated Channel Subfamily T Member 1 (KCNT1)-Related Epilepsy
Acronym: K1Te
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Collaborators: David Bearden (Unknown); University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: 992EP001
Record Dates: First submitted 2021-06-08; First posted 2021-06-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: KCNT1-Related Epilepsy
Keywords: Epilepsy of Infancy with Migrating Focal Seizures (EIMFS); Early-Onset Epileptic Encephalopathy (EOEE); Sleep-Related Hypermotor Epilepsy (SHE); Autosomal Dominant Nocturnal Frontal Lobe Epilepsy (ADNFLE)
MeSH Terms: conditions — Autosomal Dominant Nocturnal Frontal Lobe Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- EIMFS and EOEE (Up to 2 years): Participants who have been diagnosed with epilepsy of infancy with migrating focal seizures (EIMFS) and early-onset epileptic encephalopathy (EOEE) with duration of symptoms for up to 2 years will be enrolled.
  Interventions: Other: No Intervention
- EIMFS and EOEE (More than 2 years): Participants who have been diagnosed with EIMFS and EOEE with duration of symptoms for more than 2 years will be enrolled.
  Interventions: Other: No Intervention
- SHE (Up to 2 years): Participants who have been diagnosed with sleep-related hypermotor epilepsy (SHE) with duration of symptoms for up to 2 years will be enrolled.
  Interventions: Other: No Intervention
- SHE (More than 2 years): Participants who have been diagnosed with SHE with duration of symptoms for more than 2 years will be enrolled.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Administered as specified in the treatment arm.

SUMMARY:
The primary objective of the study is to characterize seizures in participants with KCNT1-related epilepsy. The secondary objectives are to characterize head growth, symptom severity, neurocognitive and social functions, adaptive behavior, sleep, quality of life, caregiver burden, and mood in participants with KCNT1-related epilepsy.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have clinically and genetically confirmed diagnosis of KCNT1-related epilepsy provided by the investigator. For purposes of this study, mutations that are genetically confirmed to cause KCNT1-related epilepsy are defined to specifically exclude known benign variants (e.g., distal C terminus, splice site, etc.).
* Willingness of the participant and/or the participant's legally authorized representative (LAR) to comply with scheduled visits and study procedures.

Key Exclusion Criteria:

* Any condition that may interfere with the assessment of KCNT1-related epilepsy and that is clearly not related to this disease (in the judgment of the investigator).
* History of human immunodeficiency virus infection.
* History of central nervous system (CNS) tumors or malignancies, including CNS metastatic disease.
* Current enrollment or past enrollment in an interventional clinical study in which an investigational gene therapy is/was administered.
* Enrollment in an interventional clinical study in which an investigational small molecule, antibody or antisense oligonucleotide (ASO) treatment or approved small molecule, antibody or ASO therapy for investigational use is administered within 1 month (or 5 half-lives of study agent, whichever is longer) prior to the screening visit.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 0 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population include participants with KCNT1-related epilepsy.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Number of Seizures in Participants with KCNT1-Related Epilepsy, Assessed by Type | Up to Month 12
  Frequency and type of seizures as recorded daily by participants (or their caregivers/observers) in an electronic seizure diary.

SECONDARY OUTCOMES:
Change from Baseline in Head Circumference | Up to Month 12
  Head circumference will be measured in participants under 18 years of age.
Clinical Global Impression-Severity (CGI-S) Scale Scores | Up to Month 12
  The CGI-S consists of a single 7-point rating score of illness severity. Raters select one response based on the following question: "Considering your total clinical experience with this particular population, how mentally ill is your participant at this time?" Scores are as follows: 1, normal, not ill at all; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill and 7, among the most severely ill participants. Higher scores indicate greater severity.
Clinical Global Impression-Change (CGI-C) Scale Scores | Up to Month 12
  The CGIC scale is a 7-point scale that requires the clinician to assess how much the participant's illness has changed relative to a baseline state at the beginning of the intervention, where 1, much better; 2, moderately better; 3, a little better; 4, the same; 5, a little worse; 6, moderately worse; 7, much worse. Higher rating will indicate worsening of the condition.
Participant-Specific Visual Analog Scale (VAS) for Most Concerning Symptoms Scores | Up to Month 12
  The participant-specific VAS for most concerning symptoms is a quality of life measurement that will be evaluated for the specified time periods. Participants report how they feel on a scale of 0 to 100, where 0 indicates being "poor" and 100 being "excellent." Up to 4 of the participant's most concerning symptoms will be assessed.
Vineland Adaptive Behavior Scales-Third Edition (Vineland-3) Composite Scores | Up to Month 12
  The Vineland-3 measures the personal and social skills of individuals from birth through adulthood. It includes 4 domains (communication, daily living skills, socialization, and motor skills) and 11 subdomains (3 each for communication, daily living skills, socialization and 2 for motor skills). Domain score ranges are as follows: 20 to 140, where 130-140, high; 115-129, moderately high; 86-114, adequate; 71-85, moderately low; 20-70, low. Composite scores are computed for each domain.
Vineland-3 Domain Scores | Up to Month 12
  The Vineland-3 measures the personal and social skills of individuals from birth through adulthood. It includes 4 domains (communication, daily living skills, socialization, and motor skills) and 11 subdomains (3 each for communication, daily living skills, socialization and 2 for motor skills). Domain score ranges are as follows: 20 to 140, where 130-140, high; 115-129, moderately high; 86-114, adequate; 71-85, moderately low; 20-70, low.
Vineland-3 Subdomain Scores | Up to Month 12
  The Vineland-3 measures the personal and social skills of individuals from birth through adulthood. It includes 4 domains (communication, daily living skills, socialization, and motor skills) and 11 subdomains (3 each for communication, daily living skills, socialization and 2 for motor skills). Subdomain score ranges from 1 to 24, where 21-24, high; 18-20, moderately high; 13-17, adequate; 10-12, moderately low and 1-9, low.
Assessment of Sleep Diary Features | Up to Month 12
  Sleep features, including total sleep time, time in bed and sleep latency. Sleep latency is defined as the amount of time taken to fall asleep after the lights have been turned off.
Number of Awakenings During Sleep | Up to Month 12
Brief Infant Sleep Questionnaire-Revised (BISQ-R) Total Scores | Up to Month 12
  BISQ-R is an age-based, norm-referenced scoring system that provides a comprehensive assessment of infant and toddler sleep patterns. It includes 3 subscales: infant sleep (IS), parent perception (PP) and parent behavior (PB). Total score ranging from 0-100 is calculated as an average of IS, PP and PB subscale scores. Higher scores denote better sleep quality, more positive perceptions of sleep quality, and parental habits that promote healthy sleep behaviors and independent infant sleep, respectively.
BISQ-R Subscale Scores | Up to Month 12
  BISQ-R is an age-based, norm-referenced scoring system that provides a comprehensive assessment of infant and toddler sleep patterns. It includes 3 subscales: IS, PP and PB. IS consists of 5 items related to sleep onset latency, number, and duration of night waking, longest stretch of sleep and total night sleep. PP consists of 3 items related to bedtime difficulty, overnight sleep, and overall child sleep problems. PB consisting of 11 items related to bedtime routine consistency, bedtime, parental behavior at time of sleep onset and night waking, sleep locations at time of sleep onset and following night waking that may impact sleep outcomes. Score ranging from 0-100 is derived for each sub-scale, with higher scores denoting better sleep quality, more positive perceptions of sleep quality, and parental habits that promote healthy sleep behaviors and independent infant sleep, respectively.
Children's Sleep Habits Questionnaire (CSHQ) Total Scores | Up to Month 12
  CSHQ is a parental report sleep screening instrument designed for preschool- and school-aged children. The scale yields both a total score and 8 subscales reflecting the following sleep domains: bedtime resistance, sleep onset delay, sleep duration, sleep anxiety, night wakings, parasomnias, sleep-disordered breathing, daytime sleepiness. Total score range between 33 and 99, with higher numbers representing more sleep problems.
CSHQ Subscale Scores | Up to Month 12
  CSHQ is a parental report sleep screening instrument designed for preschool- and school-aged children. The scale yields both a total score and 8 subscales reflecting the following sleep domains: bedtime resistance, sleep onset delay, sleep duration, sleep anxiety, night wakings, parasomnias, sleep-disordered breathing, daytime sleepiness. Score derived from each subscale range between 33 and 99, for bedtime resistance subscale, 6-18; for sleep onset/delay, 1-3; for sleep duration, 3-9; for sleep anxiety, 4-12; For night wakings, 3-9; for parasomnias, 7-21; for sleep-disordered breathing, 3-9; for daytime sleepiness, 8-24. For both total and subscale scores, higher values represent a worse outcome.
Pittsburgh Sleep Quality Index (PSQI) Total Scores | Up to Month 12
  The PSQI is a self-report questionnaire that assesses sleep quality over a 1-month time interval. It consists of 7 component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction, each of which can range from 0 to 3. The 7 components scores are then added to yield a global PSQI score in the range of 0 to 21. The higher score indicates worse sleep quality.
PSQI Subscale Scores | Up to Month 12
  The PSQI is a self-report questionnaire that assesses sleep quality over a 1-month time interval. It consists of 7 component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction, each of which can range from 0 to 3. The higher score indicates worse sleep quality.
Pediatric Quality of Life (PedsQL) Infant Scale Scores | Up to Month 12
  The PedsQL consists of 22 items comprising five dimensions: impact, cognitive functioning, sleep/rest, executive functioning, and mood/behavior that measures health related quality of life. The questionnaire asks how much of a problem each item has been during the past month. Each item is answered on a scale of 0 (never) to 4 (almost always) then the scores are transformed to a 0 to 100 scale, so that higher scores indicate better heath related quality of life.
PedsQL Core Scale Scores | Up to Month 12
  The PedsQL consists of 23 items in four generic score scales: physical functioning, emotional functioning, social functioning, and school functioning that measures health related quality of life. The questionnaire asks how much of a problem each item has been during the past month. Each item is answered on a scale of 0 (never) to 4 (almost always) then the scores are transformed to a 0 to 100 scale, so that higher scores indicate better heath related quality of life.
PedsQL Family Impact Module Scores | Up to Month 12
  The PedsQL consists of 36 items in eight dimensions: physical functioning, emotional functioning, social functioning, cognitive functioning, communication, worry, daily activities and family relationships that measures health related quality of life. The questionnaire asks how much of a problem each item has been during the past month. Each item is answered on a scale of 0 (never) to 4 (almost always) then the scores are transformed to a 0 to 100 scale, so that higher scores indicate better heath related quality of life.
Child Behavior Checklist for Ages 1.5 to 5-Language Development Survey (CBCL/1.5-5-LDS) Score | Up to Month 12
  LDS for ages of 18 months to 35 months is an important feature of the CBCL/1.5-5 which uses parent's reports to assess children's expressive vocabularies and word combinations, as well as risk factors for language delays. The LDS indicates whether a child's vocabulary and word combinations are delayed relative to norms for ages 18-35 months. The LDS can be completed for language-delayed older children for comparison with norms up to 35 months. Raw scores range from 0 to 310 words, more words is better, which are converted to a percentile ranking for gender/age based on normative data.
Child Behavior Checklist for Ages 6 to 18 (CBCL/6-18) Scores | Up to Month 12
  The CBCL/6-18 is aimed at assessing psychological adjustment and behavioral functioning of children, as rated by parents. This instrument provides a total score, an internalizing score and an externalizing score, together with 8 syndrome scale scores and 6 - Diagnostic and Statistical Manual of Mental Disorders (DSM)- oriented scale scores. It contains 113 items. Raw scores of the Total Problems Scale range from 0 to 226. Higher scores mean a worse outcome.
Adult Self-Report (ASR) Scores | Up to Month 12
  The ASR is a 126-item self-report questionnaire for adults assessing aspects of adaptive functioning and problems. The questionnaire provides scores for the following syndrome scales: anxious/depressed, withdrawn, somatic complaints, thought problems, attention problems, aggressive behavior, rule-breaking behavior, and intrusive behavior. The questionnaire provides scores for the following DSM-oriented scales: depressive problems, anxiety problems, somatic problems, avoidant personality problems, attention deficit/ hyperactivity problems (inattention and hyperactivity/impulsivity subscales), and antisocial personality problems. Additionally, the questionnaire asks about use of the following substances: tobacco, alcohol, and drugs. Items are rated on a 3-point scale: 0, not true; 1, somewhat or sometimes true; 2, very true or often true. Raw scores of the total problems scale range from 0 to 252. Higher scores mean a worse outcome.
Screen for Child Anxiety Related Emotional Disorders (SCARED)-Parent About Child Version Score | Up to Month 12
  The SCARED measures anxiety in children on a scale of 0 to 82, such that lower scores indicate low levels of anxiety, and high scores indicated high levels of anxiety.
Screen for Adult Anxiety Related Disorders (SCAARED)-Adult Version Scores | Up to Month 12
  The SCAARED measures anxiety in adults on a scale of 0 to 88 such that lower scores indicate lower levels of anxiety and high scores indicates higher levels of anxiety.
Questionnaire for Psychotic Experiences (QPE) Screening Version Scores | Up to Month 12
  The QPE is a questionnaire that is designed to quantify range of psychotic experiences, focusing on hallucinations and delusions. The 13-item screening version of the QPE that assesses the presence or absence of hallucinations and delusions will be used. Raw scores range from 0 to 26, with higher scores indicating more total and more recent symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/